CLINICAL TRIAL: NCT03957707
Title: Sterotactic Operation Integrating With Thrombolysis in Basal Ganglion Hemorrhage Evacuation: a Randomized Controlled Trial.
Brief Title: Sterotactic Operation Integrating With Thrombolysis in Basal Ganglion Hemorrhage Evacuation
Acronym: SOITBE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Ningbo No. 1 Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Second Affiliated Hospital of Wenzhou Medical University (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Zhuji People's Hospital of Zhejiang Province (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Jinhua Central Hospital (Other); Huzhou Central Hospital (Other); People's Hospital of Quzhou (Other); The Sixth Affiliated Hospital of Wenzhou Medical University (Other); The Second Affiliated Hospital of Jiaxing University (Other); Xiaoshan Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-222
Record Dates: First submitted 2019-05-19; First posted 2019-05-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Basal Ganglia Haematoma
Keywords: basal ganglion hemorrhage; stereotactic surgery; thrombolysis
MeSH Terms: conditions — Basal Ganglia Hemorrhage | interventions — Fibrinolytic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stereotactic surgery with drugs treatment (Experimental)
  Interventions: Procedure: stereotactic surgery plus thrombolysis
- drugs treatment alone (Sham Comparator)
  Interventions: Procedure: stereotactic surgery plus thrombolysis

INTERVENTIONS:
Procedure: stereotactic surgery plus thrombolysis — stereotactic puncture and aspiration to evacuate basal ganglion hematoma with or without thrombolytic agent

SUMMARY:
Spontaneous cerebral hemorrhage is one of the main causes of death and disability all over the world, accounting for 20%-30% of all cerebrovascular diseases. Minimally invasive surgery of cerebral hemorrhage, especially puncture aspiration, can improve early and long-term neurological recovery in patients with cerebral hemorrhage. Until now, no standardized practice for minimally invasive surgery of spontaneous cerebral hemorrhage has been established. Hematoma puncture and drainage based on CT scans without precise localization and personalized approach design, which may lead to poor efficacy and high risk of complications. Our hospital has much experience in treating cerebral hemorrhage with stereotactic puncture and aspiration. So we conduct a prospective multicenter randomized controlled clinical trial to determine the therapeutic effects of puncture aspiration plus thrombolysis treatment for the perioperative and long-term recovery of patients with small to moderate hematoma in deep basal ganglia via computerized precision coordinates and personalized approach design.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of spontaneous basal ganglia hemorrhage by imaging (CT, CTA, etc.) with a volume < 30 mL calculated by ABC/2 formula and Glasgow Coma Scale score ≥ 9.
2. With dysfunction such as hematoma-related motor aphasia, sensory aphasia, hemiplegic limb muscle strength ≤ grade 3 or NIHSS score ≥ 15 points.
3. Hematoma stability shown by a CT scan at least 6 hours after the diagnostic CT (hematoma volume increase < 5 ml by ABC/2 formula)
4. Diagnostic CT scan should be obtained within 24 hours after the onset of symptoms. Cases with unclear onset time should be excluded.
5. Randomization within 72 hours after diagnostic CT.
6. Surgery should be performed within 72 hours after onset.
7. SBP <180 mmHg maintained for 6 hours prior to randomization.
8. Age between 18-70 years old.
9. mRS score ≤ 1 in past medical history.
10. Patients who are suitable and willing to be randomized to "puncture aspiration + urokinase" or conservative medical treatment.

Exclusion Criteria:

1. Hematoma involves other structures such as the thalamus and midbrain.
2. Mass effect or hydrocephalus due to intraventricular hemorrhage.
3. Imaging-based diagnosis of cerebrovascular abnormalities such as ruptured aneurysm, arteriovenous malformation (AVM) and moyamoya disease as well as hemorrhagic transformation of ischemic infarct and recent recurrence (within 1 year) of cerebral hemorrhage.
4. Manifestation of early stage cerebral herniation such as ipsilateral pupil changes and midline shift exceeding 1 cm.
5. Patients with unsteady hematoma or with progression to intracranial hypertension syndrome.
6. Patients with any irreversible coagulopathy or known coagulation disorders; platelet count <100,000; INR > 1.4.
7. Patients requiring long-term use of anticoagulants.
8. Patients taking dabigatran, apixaban and/or rivaroxaban (or similar drugs of the same category) before symptoms arise.
9. Bleeding in other sites, including retroperitoneal, gastrointestinal, genitourinary or respiratory tract bleeding; superficial or skin surface bleeding mainly occurring in the vascular puncture site or transvenous approach (eg. arterial puncture, venous incision, etc. ) or in the recent surgical site.
10. May be pregnant in the near future or already pregnant.
11. Previously enrolled in this study.
12. Participating in other interventional medical research or clinical trials at the same time.

    Patients enrolled in observational, natural history and/or epidemiological studies (without intervention) are eligible for this trial.
13. Patients with an expected survival of less than 6 months.
14. Patients with severe co-morbidity (including hepatic, renal, gastrointestinal, respiratory, cardiovascular, endocrine, immune and/or hematological disorders) which may affect the outcome assessment.
15. Patients with mechanical heart valve. Biological valves are acceptable.
16. Patients with risk of embolism (including a history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis or subacute bacterial endocarditis). Atrial fibrillation without mitral stenosis is acceptable.
17. Investigators believe co-morbidities would be detrimental to the patient when the study begins.
18. Patients difficult to follow up or with poor compliance due to various reasons (such as geographical and social factors, drug or alcohol abuse, etc.)
19. Patient or his or her legal guardian/representative is unable or unwilling to give the written informed consent.
20. Patients is in a condition that is not suitable for "puncture aspiration + urokinase" treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Favorable Functional Outcome as Defined by the modified Rankin Scale (mRS) Score | 6 months
  Functional independence is defined as achieving a score of 0, 1, or 2 on the mRS. The mRS is a 7-point scale that measures the degree of disability or dependence in the daily activities of patients who have had a stroke. The scale ranges from 0 (no symptoms) to 6 (dead).

SECONDARY OUTCOMES:
All-Cause Mortality | 6 months
Change in Barthel Index (BI) | 6 months
  Functional status in activities of daily living (ADL) will be assessed using the Barthel Index (BI). The BI score ranges from 0 (completely dependent) to 100 (fully independent).
Changes in Glasgow Outcome Scale-Extended (GOS-E) score | 6 months
  The GOS-E is an 8-point scale that categorizes global outcomes from Dead (1) to Upper Good Recovery (8).
Hematoma clearance rate | 1 day and one month
Total duration of the initial hospital stays | one month
Total direct medical costs during the index hospitalization | one month

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided